CLINICAL TRIAL: NCT00346905
Title: Endoscopic Implantation of Enteryx for the Treatment of Gastroesophageal Reflux Disease (GERD): Post Market Study
Brief Title: Endoscopic Implantation of Enteryx for the Treatment of GERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Douglas Pleskow, Associate Clinical Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003P000277
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD; Gastroesophageal Reflux Disease; Reflux; Enteryx
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — ethylene-vinyl alcohol copolymer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Those receiving Enteryx treatment
  Interventions: Drug: Enteryx

INTERVENTIONS:
Drug: Enteryx

SUMMARY:
The study objective is to assess the long term safety and effectiveness of Enteryx device in commercial use. The long-term effects beyond one year of treatment with Enteryx have not been established.

DETAILED DESCRIPTION:
The Enteryx procedure kit is indicated for endoscopic injection into the region of the lower esophageal sphincter (LES) for the treatment of symptoms due to gastroesophageal reflux disease (GERD) symptoms in patients responding to and requiring daily pharmacological therapy with proton pump inhibitors (PPI's).

The study design consists of two parts, Part A and Part B. Part A will enroll patients who received Enteryx treatments after approval and Part B will enroll patients previously enrolled and treated in the IDE study #G000065. In total there will be at least 300 patients enrolled in Part A and Part B with 36 months of follow-up Part A: Approximately 150 to 200 patients will be enrolled from 22 centers. After patients have determined with their physicians that Enteryx is an appropriate course of therapy for their GERD symptoms, they will be asked to participate in this trial. Patients will be followed for adverse events, medication use, and GERD-HRQL symptoms at baseline, day of treatment, one month, six months, twelve months, twenty-four months, and thirty-six months. The final study visit will be thirty-six months after the last Enteryx injection. In addition, all Part A patients will be contacted by the Site at least quarterly to obtain current adverse event information. This adverse event information will be solicited from the Site by the Sponsor at least quarterly. Part B: All US IDE patients (approximately 150 patients) will be asked to enroll. Patients will be followed for adverse events, medication use, and GERD-HRQL symptoms at two visits beyond the follow-up prescribed in the IDE study, namely 24 and 36 months after the last Enteryx injection received in the IDE study. Parts A and B: There will be a breakdown of adverse events based on retreatment status. Any subsequent procedures or interventions related to GERD or Enteryx, whether surgical (such as fundoplication) or non-surgical (such as an alternative endoscopic treatment for GERD), will be collected and reported.

H0: (Null hypothesis): Proportion of patients exhibiting clinically significant improvement in reduction of PPI therapy ≤ 0.5

Ha: (Alt. hypothesis): Proportion of patients exhibiting clinically significant improvement in reduction of PPI therapy > 0.5

The Sponsor will examine the proportion of patients who have clinically significant reduction in PPI therapy at the 12, 24 and 36 month follow-ups, in an identical manner to that used for the patients in the IDE trial. The "clinically significant reduction" is defined as either elimination of medication use or reduction in dosage of ≥50%. The criterion for success is defined as more than half of patients demonstrating this degree of medication reduction. The hypothesis is tested by p-value and construction of the exact 95% Clopper-Pearson confidence intervals around the observed proportion of patients who meet the criterion for success. The longitudinal post-procedure follow-up data across time (repeated measures) will be analyzed to determine patterns and trends for all primary endpoints. The hypothesis stated above will also be evaluated in the subset of patients that underwent retreatment prior to amendment v.14Oct05.

ELIGIBILITY:
Inclusion Criteria:

* GERD responsive to and requiring daily PPI therapy

Exclusion Criteria:

* Esophageal varices, particularly related to portal hypertension • Patients whom the physician determines to be a poor candidate for endoscopic procedures and/or anesthesia.

Patients must also be willing to allow their data to be shared with the Sponsor and FDA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Chen, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Referral patients experiencing moderate to severe GERD
Pre-assignment Details: Those not meeting inclusion/exclustion criteria were not included
Groups:
- Group 1: Patients that are GERD responsive and requiring daily PPI therapy
Period: Overall Study
Arm/Group | Group 1
Started | 16
Completed | 12
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Patients experiencing moderate GERD
Arm/Group | Group 1
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants] — Participants analyzed are over 18 years of age.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 10
    >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Reduction of PPI Usage at 12, 24, and 36 Month Follow-ups Compared to Baseline in Both Singly Treated and Retreated Patients.
Description: Clinically significant reduction of PPI usage is defined as either elimination of medication use or reduction in dosage of ≥50% as compared to baseline. The criterion for success is defined as more than half of patients demonstrating this degree of medication reduction.
Time Frame: 3 years either baseline to 12m, baseline to 24m, baseline to 36m
Population: Overall Number of Participants Analyzed (16) will differ at 12m, 24m, and 36m intervals due to patients who were available at the given follow-up interval.
Measure: Number; unit: % of Participants
Groups:
- Enteryx Treatment: Those receiving Enteryx treatment
  Enteryx
Arm/Group | Enteryx Treatment
Number analyzed (Participants) | 16
% of Participants
  clinically significant reduction of PPI usage 12m | 56.25
  clinically significant reduction of PPI usage 24m: number analyzed (Participants) | 11
  clinically significant reduction of PPI usage 24m | 45.45
  clinically significant reduction of PPI usage 36m: number analyzed (Participants) | 12
  clinically significant reduction of PPI usage 36m | 50.00

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Group 1 - Single Arm: Those experiencing GERD
Arm/Group | Group 1 - Single Arm
Serious Adverse Events (participants affected / at risk) | 10/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Single Arm (N=16)
Flutter Fibrillation (Cardiac disorders) | 1 (1)
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Retrosternal Chest Pain (General disorders) | 1 (1)
Severe Chest Pain / Myocardial Infarction (Cardiac disorders) | 1 (1)
Malignant Nodule in Thyroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chemical Mediastinitis (Infections and infestations) | 1 (1)
Pleuritic Chest Pain with Inspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Torn Rotator Cuff (Musculoskeletal and connective tissue disorders) | 1 (1)
Hiatal Hernia Repair (Surgical and medical procedures) | 1 (1)
Nissen Fundoplication for Severe GERD (Gastrointestinal disorders) | 1 (1)
Bleeding Esophageal Ulcer (Gastrointestinal disorders) | 1 (1)
Chest Pain secondary to Coronary Artery Disease (Cardiac disorders) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rigors "Shaking Chills" (General disorders) | 1 (1)
C-Diff Colitis (Infections and infestations) | 1 (1)
Heart Attack (Cardiac disorders) | 1 (1)
Nissen Fundoplication Repair with Hospital Stay for GERD and Pulmonary Symptoms (Surgical and medical procedures) | 1 (1)
Nissen Fundoplication for GERD. Hospitalized for 2 days post surgery. (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Single Arm (N=16)
Worse Than Ever Heartburn. Woke Pt. from Sleep. (Gastrointestinal disorders) | 1 (1)
Herniated Cervical Disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 6 (7)
Arthritic low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in the middle of Chest brought on by physical activity (General disorders) | 1 (1)
Retrosternal Chest Pain (General disorders) | 9 (9)
Shortness of Breath brough on by physical activity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Hiatal Hernia (Gastrointestinal disorders) | 1 (1)
Schatzski's Ring (Gastrointestinal disorders) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diverticulosis of Sigmoid Colon (Gastrointestinal disorders) | 1 (1)
Excessive Gas (Gastrointestinal disorders) | 1 (1)
Patient with complaint of left lateral wall discomfort in left axilla. Occasional/short lasting (General disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Low grade fever (General disorders) | 1 (1)
Minor Cold (Infections and infestations) | 1 (1)
More servere hearburn than Baseline (Gastrointestinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Burping (Gastrointestinal disorders) | 1 (1)
Sinusitis with asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Worsening of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bleeding gastric ulcer (Gastrointestinal disorders) | 1 (2)
Exacerbation of reflux due to medication taken for pneumonia (Gastrointestinal disorders) | 1 (1)
Gastric fistula (Gastrointestinal disorders) | 1 (1)
High Blood Pressure (Vascular disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Viral illness accompanied by headache, nauseau, and vomiting (Infections and infestations) | 1 (1)
Torn ligmament in left shoulder (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Cold like symtoms (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Exacerbated GERD symptoms - gagging, coughing, mucus due to stress when patient's mother was ill. (Gastrointestinal disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Worsening of GERD Symptoms (Gastrointestinal disorders) | 2 (2)
More severe heartburn than baseline (Gastrointestinal disorders) | 1 (1)
Exacerbation of GERD symptoms similar to baseline (Gastrointestinal disorders) | 1 (1)
Increase in severity of nausea (Gastrointestinal disorders) | 1 (1)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased Burping (Gastrointestinal disorders) | 1 (1)
Mild Retrosternal Chest Pain (General disorders) | 1 (1)
Difficulty Swallowing (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Trouble Swallowing (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No